CLINICAL TRIAL: NCT00355277
Title: Local Anaesthetic Effects of Transcutaneous Amitriptyline in Human Volunteers : a Controlled, Double-blinded, Randomised Study Versus Placebo and Transcutaneous Local Anaesthetic (EMLA(R))
Brief Title: Local Anaesthetic Effects of Transcutaneous Amitriptyline
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU63-0014
Record Dates: First submitted 2006-07-20; First posted 2006-07-21 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Healthy Volunteers
Keywords: Tricyclic antidepressants; Neuropathic pain; Local anaesthesia; Transcutaneous
MeSH Terms: conditions — Neuralgia | interventions — Amitriptyline

INTERVENTIONS:
Drug: Amitriptyline

SUMMARY:
The aim of this study is to assess the local anaesthetic effects of amitriptyline applied on the skin of human volunteers, considering the differential effects on mechanic and thermic sensitivity, the local and general tolerance, and the systemic absorption of the drug. The solution used for dilution of amitriptyline is the only one known to allow transcutaneous absorption of the drug [1]. Considering that the peripheral sensitive fibre is a possible site of action of tricyclic antidepressants for relieving neuropathic pain [2,3], this is a first step study before further assessment of the therapeutic effects of transcutaneous amitriptyline.

DETAILED DESCRIPTION:
Sixteen male healthy volunteers are enrolled for this study. They receive in a randomised order on six regions of dorsal skin (after previous targetting by ink marks) the six following treatments : lidocaïne-prilocaïne anaesthetic cream (EMLA (R)), normal saline, amityptiline hydrochloride diluted in solution of water (%), isopropanol (%) , glycerol (%), titrated with sodium hydroxide for pH=8.5, at four different concentrations (0,25, 50 and 100 mM). The person in charge of local application does not participate to further examination. Immediately after one hour of application, the volunteer is examined, and then every 2 hours during 8 hours, and 24 hours after the end if application. Every trial includes, for every treated area, (a) measurement of sensitive and nociceptive threshold to Von Frey hair application, (b) assessment of sensation induced by cold and heat after Rolltemp TM application, (c) measurement of sensitive threshold to cold, then sensitive and nociceptive thresholds to heat with Thermotest TM, (d) clinical evaluation of tolerance to the treatment, (e) blood sampling for measuring amitriptylinemia (HPLC). The possible residual anaesthetic effects of the treatment are assessed one and three weeks after the application, by measurement of sensitive and nociceptive threshold to Von Frey hair application. The statistical analysis will use two-way ANOVA, considering the following factors : treatment, time, order, subject, subject/order.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* history of intolerance to amitriptyline, lidocaine or prilocaine
* cardiac predisposition to intolerance to tricyclic antidepressants

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16
Dates: Start 2005-11; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Claude DUBRAY, Pr, Principal Investigator — CENTRE DE PHARMACOLOGIE CLINIQUE; Christian DUALE, Dr, Study Director — CENTRE DE PHARMACOLOGIE CLINIQUE; PICKERING gisele, Dr, Study Director — CENTRE DE PHARMACOLOGIE CLINIQUE
Locations (1):
- Centre de Pharmacologie Clinique /Cic, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Background] Kissin I, McDanal J, Xavier AV. Topical lidocaine for relief of superficial pain in postherpetic neuralgia. Neurology. 1989 Aug;39(8):1132-3. doi: 10.1212/wnl.39.8.1132-a. No abstract available. PMID 2761713
- [Background] Sawynok J, Esser MJ, Reid AR. Antidepressants as analgesics: an overview of central and peripheral mechanisms of action. J Psychiatry Neurosci. 2001 Jan;26(1):21-9. PMID 11212590
- [Background] McQuay HJ, Tramer M, Nye BA, Carroll D, Wiffen PJ, Moore RA. A systematic review of antidepressants in neuropathic pain. Pain. 1996 Dec;68(2-3):217-27. doi: 10.1016/s0304-3959(96)03140-5. PMID 9121808
- [Result] Duale C, Daveau J, Cardot JM, Boyer-Grand A, Schoeffler P, Dubray C. Cutaneous amitriptyline in human volunteers: differential effects on the components of sensory information. Anesthesiology. 2008 Apr;108(4):714-21. doi: 10.1097/ALN.0b013e3181672632. PMID 18362604
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/18362604